CLINICAL TRIAL: NCT00456027
Title: A Placebo-Controlled Study to Investigate the Impact of Diamyd® on the Diabetes Status of Patients With LADA (Latent Autoimmune Diabetes in Adult)
Brief Title: Safety of Diamyd® in Patients With LADA (Latent Autoimmune Diabetes in Adult)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Diamyd Therapeutics AB (Industry)
Responsible Party: Managing Director, Diamyd Therapeutics AB
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D/P2/04/2; EUDRACT 2004-001998-25
Record Dates: First submitted 2007-04-03; First posted 2007-04-04 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2007-04

CONDITIONS: Latent Autoimmune Diabetes in Adult (LADA)
Keywords: Type 2 Diabetes; LADA; Latent Autoimmune Diabetes in Adult; Autoimmunity; HbA1c; C-peptide
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Autoimmune Diseases | interventions — Aluminum Hydroxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: rhGAD65 formulated in Alhydrogel® (Diamyd®) — 20 micrograms of rhGAD65 formulated in Alhydrogel® administered subcutaneously twice 4 weeks apart

SUMMARY:
This is a study to investigate the safety of 20ug Diamyd® (rhGAD65 formulated in Alhydrogel®), administered subcutaneously four weeks apart in patients with Latent Autoimmune Diabetes in Adult (LADA).

ELIGIBILITY:
Key Inclusion Criteria:

* Male and female patients between 30-70 years of age diagnosed with type 2 diabetes within 5 years
* Presence of GAD65 antibodies
* Detectable C-peptide level
* Patients requiring treatment with diet and/or oral hypoglycaemic agents (OHA)
* Written informed Consent

Key Exclusion Criteria:

* Treatment with insulin
* Intolerance to OHA
* Secondary diabetes mellitus
* History of certain diseases or conditions (e.g. anaemia, epilepsy, head trauma, neurological disease, alcohol or drug abuse, HIV, hepatitis)
* Treatment with any vaccine within one month prior to first Diamyd® dose or planned treatment with vaccine up to 2 months after the second Diamyd® dose
* Participation in other clinical trials with a new chemical entity within the previous 3 months
* Pregnancy (or planned pregnancy within one year after 2nd administration)
* Presence of associated serious disease or condition which in the opinion of the investigator makes the patient non-eligible for the study
* Significant illness other than diabetes within 2 weeks prior to first dosing
* Unwillingness to comply with the provisions of the protocol
* Clinically significant history of acute reaction to drugs in the past
* Treatment with immunosuppressants

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2004-12; Primary Completion 2008-03 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
The development over time of safety variables, i.e. injection site discomfort, vital signs, laboratory values and AEs/SAEs as well as development of diabetes status, i.e. HbA1c, C-peptide, blood glucose and insulin requirement. | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Carl-David Agardh, MD, phD, Principal Investigator — University Hospital MAS, Malmö, Sweden
Locations (17):
- Sweden (17):
  - Alingsås Hospital, Alingsås
  - Falu Hospital, Falun
  - Capio Lundby Hospital, Gothenburg
  - Härnösand Hospital, Härnösand
  - Helsingborg Hospital, Helsingborg
  - Karlstad Central Hospital, Karlstad
  - Central Hospital, Kristianstad, Kristianstad
  - Sunderby Hospital, Luleå
  - University Hospital MAS, Malmo
  - Vrinnevi Hospital, Norrköping
  - Odensala Health Clinic, Östersund
  - Skellefteå Hospital, Skellefteå
  - S:t Göran Hospital, Stockholm
  - Stockholm South General Hospital, Stockholm
  - Norrlands University Hospital, Umeå
  - Uppsala University Hospital, Uppsala
  - Växjö Central Hospital, Vaxjo